CLINICAL TRIAL: NCT01494740
Title: Immunogenicity and Safety of an Inactivated Split-virion 2009 Pandemic Influenza A H1N1 Vaccine in Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SIBP-2009-1
Record Dates: First submitted 2011-12-15; First posted 2011-12-19 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2009-10

CONDITIONS: Influenza
Keywords: H1N1; Vaccine; Immunogenicity; Safety; infants
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- split-virion, non-adjuvanted vaccine of 7.5 μg (Experimental): split-virion, non-adjuvanted H1N1 vaccine of 7.5 μg.
  Interventions: Biological: split-virion, non-adjuvanted vaccine of 7.5 μg
- split-virion, non-adjuvanted vaccine of 15 μg (Experimental): split-virion, non-adjuvanted H1N1 vaccine of 15 μg.
  Interventions: Biological: split-virion, non-adjuvanted H1N1 vaccine of 15 μg
- split-virion, non-adjuvanted vaccine of seasonal influenza (Placebo Comparator): split-virion, non-adjuvanted H1N1 vaccine of seasonal influenza.
  Interventions: Biological: split-virion, non-adjuvanted vaccine of seasonal influenza

INTERVENTIONS:
Biological: split-virion, non-adjuvanted vaccine of 7.5 μg — 120 infants were assigned to receive 2 dose of 7.5μg split-virion, non-adjuvanted H1N1 vaccine.
  Arms: split-virion, non-adjuvanted vaccine of 7.5 μg
Biological: split-virion, non-adjuvanted H1N1 vaccine of 15 μg — 120 infants were assigned to receive 2 dose of 15μg split-virion, non-adjuvanted H1N1 vaccine.
  Arms: split-virion, non-adjuvanted vaccine of 15 μg
Biological: split-virion, non-adjuvanted vaccine of seasonal influenza — 120 infants were assigned to receive 2 dose of split-virion, non-adjuvanted seasonal influenza vaccine.
  Arms: split-virion, non-adjuvanted vaccine of seasonal influenza

SUMMARY:
The aim of this study is to investigate the immunogenicity and safety of the inactivated split-virion vaccine in infants.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants aged between 6 and 35 months
2. full-term birth with birth weight above 2,500 grams
3. Subject and parent/legal representative should be present at all scheduled visits and to obey all trial procedures

Exclusion Criteria:

1. Volunteers in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the first trial vaccination
2. Volunteers allergic to ingredient of vaccine composition (can be checked from vaccination history), especially to egg
3. History of progressive or severe neurologic disorder
4. Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain
5. Known or suspected impairment/alteration of immune function, for example receiving immunosuppressive therapy or receiving blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation
6. Asthma that is unstable or required emergent care, hospitalization or intubation during the past two years or that required the use of oral or intravenous corticosteroids
7. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
8. History of thyroidectomy or thyroid disease that required medication within the past 12 months
9. Serious angioedema episodes within the previous 3 years or requiring medication in the previous two years
10. Guillain-Barre Syndrome
11. Self-reported seropositivity for Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C
12. Any other vaccines or immunoglobulin preparation within 1 weeks prior to enrollment
13. Axillary temperature ≥ 38.0 degrees Celsius within 3 days of intended study vaccination
14. Any conditions may influence the evaluation

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 312 (Actual)
Dates: Start 2009-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Hemagglutination inhibition antibody titer | Days 35

SECONDARY OUTCOMES:
Occurrence of solicited local and systemic adverse events after vaccination | Day0-42

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Provincial Center of Disease Prevention and Control Changsha, Hunan, China, Changsha, China

REFERENCES:
- [Derived] Wang S, Dong J, Chai W, Li F, Wang S, Sun B, Chen Z. Immunogenicity of a monovalent 2009 influenza A (H1N1) vaccine in infants: randomized, observer-masked, single-center clinical study. Springerplus. 2014 Jul 31;3:397. doi: 10.1186/2193-1801-3-397. eCollection 2014. PMID 25110632